CLINICAL TRIAL: NCT07316933
Title: Acute Responses to Different Blood Flow Restriction Exercise Configurations With Dynamic Pressure Compared to Fixed Pressure in Patients With Severe Gonarthrosis
Brief Title: Acute Exercise Responses With Blood Flow Restriction Under Dynamic Pressure Compared to Fixed Pressure in Patients With Severe Gonarthrosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Adrián Escriche Escuder, Assistant professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-FIS-3955989
Record Dates: First submitted 2025-12-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Severe Knee Osteoarthritis
Keywords: blood flow restriction; exercise; gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low-load resistance exercise with moderate blood occlusion and dynamic pressure. (Experimental): A single session of exercise, 30% repetition maximum, 50% blood occlusion, and dynamic pressure
  Interventions: Device: Moderate-intensity resistance exercise with low arterial occlusion pressure and dynamic pressure.
- Low-load resistance exercise with moderate blood occlusion and fixed pressure. (Experimental): A single session of exercise, 30% repetition maximum, 50% blood occlusion, and fixed pressure
  Interventions: Device: Moderate-intensity resistance exercise with low arterial occlusion pressure and fixed pressure.
- Moderate-load resistance exercise with low blood occlusion and dynamic pressure. (Experimental): A single session of exercise, 50% repetition maximum, 30% blood occlusion, and dynamic pressure
  Interventions: Device: Low-intensity resistance exercise with high arterial occlusion pressure and dynamic pressure.
- Moderate-load resistance exercise with low blood occlusion and fixed pressure. (Experimental): A single session of exercise, 50% repetition maximum, 30% blood occlusion, and fixed pressure
  Interventions: Device: Low-intensity resistance exercise with high arterial occlusion pressure and fixed pressure.
- Low-load resistance exercise with high blood occlusion and dynamic pressure (Experimental): A single session of exercise, 15% repetition maximum, 80% blood occlusion, and dynamic pressure
  Interventions: Device: Low-intensity resistance exercise with moderate arterial occlusion pressure and dynamic pressure.
- Low-load resistance exercise with high blood occlusion and fixed pressure (Experimental): A single session of exercise, 15% repetition maximum, 80% blood occlusion, and fixed pressure
  Interventions: Device: Low-intensity resistance exercise with moderate arterial occlusion pressure and fixed pressure.

INTERVENTIONS:
Device: Low-intensity resistance exercise with moderate arterial occlusion pressure and dynamic pressure. — A single quadriceps extension exercise at 30% of 1 repetition maximum (1RM) with dynamic occlusion at 50% of limb occlusion pressure (LOP), performing 4 sets of 30, 15, 15, 15 repetitions with 30 seconds of rest between sets.
  Arms: Low-load resistance exercise with high blood occlusion and dynamic pressure
Device: Low-intensity resistance exercise with moderate arterial occlusion pressure and fixed pressure. — A single quadriceps extension exercise at 30% of 1RM with fixed occlusion at 50% of limb occlusion pressure (LOP), performing 4 sets of 30, 15, 15, 15 repetitions with 30 seconds of rest between sets.
  Arms: Low-load resistance exercise with high blood occlusion and fixed pressure
Device: Moderate-intensity resistance exercise with low arterial occlusion pressure and dynamic pressure. — A single quadriceps extension exercise at 50% of 1RM with dynamic occlusion at 30% of limb occlusion pressure (LOP), performing 4 sets of 30, 15, 15, 15 repetitions with 30 seconds of rest between sets.
  Arms: Low-load resistance exercise with moderate blood occlusion and dynamic pressure.
Device: Moderate-intensity resistance exercise with low arterial occlusion pressure and fixed pressure. — A single quadriceps extension exercise at 50% of 1RM with a fixed occlusion of 30% of the limb occlusion pressure (LOP), performing 4 sets of 30, 15, 15, 15 repetitions with 30 seconds of rest between sets.
  Arms: Low-load resistance exercise with moderate blood occlusion and fixed pressure.
Device: Low-intensity resistance exercise with high arterial occlusion pressure and dynamic pressure. — A single quadriceps extension exercise at 15% of 1RM with a dynamic occlusion of 80% of the limb occlusion pressure (LOP), performing 4 sets of 30, 15, 15, 15 repetitions with 30 seconds of rest between sets.
  Arms: Moderate-load resistance exercise with low blood occlusion and dynamic pressure.
Device: Low-intensity resistance exercise with high arterial occlusion pressure and fixed pressure. — A single quadriceps extension exercise at 15% of 1RM with a fixed occlusion of 80% of the limb occlusion pressure (LOP), performing 4 sets of 30, 15, 15, 15 repetitions with 30 seconds of rest between sets.
  Arms: Moderate-load resistance exercise with low blood occlusion and fixed pressure.

SUMMARY:
This study aims to evaluate the acute effects of blood flow restriction (BFR) training on hypoalgesia and neuromuscular responses in patients with severe gonarthrosis by comparing the application of pressure with a dynamic versus a fixed configuration. There will be six different training conditions with varying levels of blood flow occlusion (%BFR) and percentage of load (%RM): 1) 30% RM and 50% BFR with dynamic pressure; 2) 30% RM and 50% BFR with fixed pressure; 3) 50% RM and 50% BFR with dynamic pressure; 4) 50% RM and 50% BFR with fixed pressure; 5) 30% RM and 80% BFR with dynamic pressure; 6) 30% RM and 80% BFR with fixed pressure.

Each participant will complete six individual sessions under different training conditions, assigned in a random order with a 72-hour interval between each session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 85 years
* Diagnosis of severe gonarthrosis according to the clinical and radiographic criteria of the American College of Rheumatology guidelines.
* On the waiting list for unilateral total knee replacement (TKR) surgery

Exclusion Criteria:

* Pain in the contralateral leg with an intensity ≥80/100 mm on the visual analog scale (VAS) during daily activities.
* Previous hip or knee replacement surgery and osteotomy within the last year.
* Autoimmune arthritis
* Medical conditions that contraindicate exercise.
* Participation in exercise programs (>2 days/week with training at intensities of 10-15 1RM) in the previous six months.
* History of stroke, brain surgery, major depression, or self-reported cognitive impairment that could affect performance in the study.
* Cardiovascular, thrombotic, or vascular risk factors (uncontrolled hypertension, peripheral arterial disease, history of deep vein thrombosis or pulmonary embolism, heart failure, severe varicose veins, or uncontrolled anticoagulant therapy).
* Skin or local alterations at the cuff application site (ulcers, open wounds, infections, lymphedema, or severe edema).
* Inability to communicate normally or with impaired communication skills.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at rest (Visual Analogue Scale, 0-10) | Periprocedural
  Pain intensity perceived on a Visual Analogue Scale, at rest, being 0 no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Pressure pain threshold | Periprocedural
  Pressure pain threshold measured in the middle deltoid (peripheral sensitivity) and tibialis anterior (central sensitivity), using an algometer
Perceived exertion scale (The BORG CR10 Scale) | Periprocedural
  The BORG CR10 Scale is a subjective tool used to measure the intensity of the perceived exertion of a person during an activity through a rate of perceived exertion (RPE). It is scored on a scale of 0 to 10, where 0 is no exertion and 10 is maximum exertion.
Surface electromyography | Periprocedural
  Surface electromyography for the study of muscle recruitment (vastus medialis and vastus lateralis)
Occurrence of adverse effects | Immediately after the intervention, 72 hours later, and two weeks after the study ended.
  Occurrence of adverse effects (e.g., pain, delayed onset muscle soreness, sudden weakness of the trained limb, redness or swelling of the trained limb, etc.) by self-report.
Kinesiophobia (The Tampa Scale for Kinesiophobia) | Baseline
  The Tampa Scale for Kinesiophobia is a questionnaire designed to assess fear of movement and avoidance of physical activity due to pain. It consists of 17 items answered on a scale of 1 (strongly disagree) to 4 (strongly agree), measuring two main factors: fear of movement and activity avoidance. The total score ranges from 17 to 68 points, with higher scores indicating greater kinesophobia.
Pain catastrophizing | Baseline
  The Pain Catastrophizing Scale includes 13 items in total (0-52 points) that describe different thoughts and feelings associated with pain. The PCS consists of 5 grades: 0 not at all, 1 a little, 2 moderately, 3 a lot, and 4 always. The participant must mark their situation for each case. Higher scores correspond to higher levels of pain catastrophizing
Functional Measure (Western Ontario and McMaster Universities Osteoarthritis Index) | Baseline
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a questionnaire designed to assess pain, stiffness, and function in patients with knee and hip osteoarthritis. It consists of 24 items, divided into three subscales that assess pain (5 items), stiffness (2 items), and physical function (17 items). Responses are given on a 0-to-4 Likert-type scale, where higher scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available from the corresponding author upon reasonable request.